CLINICAL TRIAL: NCT01750424
Title: 3-D Imaging Assessment of Scar Formation and Would Healing in Fat Grafted vs Non-Fat Grafted Facial Reconstruction Wound Sites
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIC-1209010842
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Scar Formation; Autologous Fat Grafting
Keywords: Scar; Fat Grafting; Adipose Grafting; 3-D imaging; Manchester Scar Scale
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fat Grafted (Experimental): The experimental arm of the study will be composed of 15 patients who undergo autologous fat grafting into the site of the facial reconstructive scar at 3 months post-operatively. A small amount of fat will be removed near the umbilicus through a cannula using local anesthetic and a small, 2-3mm incision just barely large enough for the cannula to pass. That fat will be injected directly under the scar site in those patients using a similar cannula, local anesthetic, and small, 2-3mm incision. No sutures will be required at either the donor or injection site. Patients will subsequently return to clinic for 3-D photographic assessment at 3, 6 and 12 months post-fat grafting. The images generated at each session will be provided to a group of assessors for evaluation. They will either use the Manchester Scar Scale or the modified Manchester Scar Scale depending on whether they are within the health care profession.
  Interventions: Procedure: Autologous Fat Grafting
- Non-fat grafted (Placebo Comparator): The control arm will be composed of 15 patients who undergo no intervention. These patients will be identified at 3 months post-operatively from their facial reconstruction. They will undergo no fat-grafting but will be followed up with the same frequency as the experimental group, at 3 months, 6 months, and 12 months after their initial 3 month post-surgical follow-up. 3-D images will be taken at each appointment and will be distributed to all assessors. Assessors will use either the Manchester Scar Scale or a modified Manchester Scar Scale to evaluate the appearance of the scar at each time point.
  Interventions: Other: No intervention

INTERVENTIONS:
Procedure: Autologous Fat Grafting
  Other Names: Fat Grafting; Adipose Grafting
  Arms: Fat Grafted
Other: No intervention — Subjects in this arm will only be followed up and have no procedure performed.
  Arms: Non-fat grafted

SUMMARY:
The purpose of this study is to assess scar-formation and wound healing following the use of autologous fat grafting in facial reconstruction patients. Patients who have undergone facial reconstruction in the last 3 months will be randomized into two groups, one receiving fat grafting and one not receiving any intervention. These patients will continue to follow-up in our clinic for one year, with 3-D images taken at each follow-up visit to assess scar formation and wound healing. Assessment of the scar will be undertaken by both healthcare personnel as well as general lay public. We hypothesize that patients undergoing fat grafting to the wound site will achieve a more aesthetically appealing result, with less scarring and improved wound healing as judged by both the general public and healthcare professionals.

DETAILED DESCRIPTION:
A variety of local and regional skin flaps are used for reconstruction of skin defects on the face with the intention of full wound closure, healing, and scar minimization. Scarring is an unavoidable consequence of wound healing, especially after significant facial reconstruction. Fibroblasts migrate to the injurious site where they proliferate and deposit collagen. The collagenous proteins serve to fill in the wound defect and allow epithelial cells to accumulate and repopulate the skin surface. The collagenous base is subsequently exchanged for various types of collagen and is crosslinked. Although scar formation is an important component of wound healing, patients develop scars differently based upon location and biology of the subject. Excessive scar formation may result from excessive collagen production and inadequate collagen remodeling (Gurtner).

Much effort has focused on minimizing scar formation. Such techniques have included rigorous sterilization techniques, smaller, more linear incisions, and incisions that follow normal tension lines in the skin to name only a few. However, these techniques have been mostly limited to intraoperative or pre-operative measures. And while successful in minimizing scar burden, these techniques do not address scar management post operatively.

Wound healing and scar formation follow complex biological processes dependent on inflammatory cells and growth factors. It has been shown in utero that fetal wounds are capable of scarless healing during a phase of gestation when wounds heal with a paucity of inflammatory cells (Soo, Frantz). This principle was further studied in immune deficient mice lacking both macrophages and neutrophils, which are critical to the inflammatory response. Within this experiment, both groups of mice (immunodeficient and normal mice) healed the wounds, the immunodeficient mice did so in a scarless manner (Mori, Martin). Extrapolating this information to current surgical patients, the development of an immunomodulating measure is critical to inhibiting and managing scar formation.

Adipose derived mesenchymal stem cells (ADSCs) have been studied with regard to their role in the wound healing and scar formation process and have shown great promise. In experimental studies, ADSCs have shown to promote angiogenesis, granulation and reepithelialization of the overlying wound (Ebrahimian). Whether directly or indirectly through these processes, the ADSCs also improve the appearance of resultant scars by decreasing size, contrast of scar color, and improving pliability of the scar (Blanton, Yun). However, it is not to be confused that all adipose tissue is equivalent with ADSCs. Rather, ADSCs are a particular line of cells found within adipose tissue that have the unique capability of differentiating into a variety of types of tissues, from bone to cartilage to further adipose tissue (Zuk). These cells are capable of being harvested and cultured from adipose tissue within subjects and then subsequently injected into the wound site of interest.

Fat grafting is a similar but less involved technique that harvests autologous adipose tissue but does not use cell culture techniques to isolate ADSCs from other cell lineages. Fat grafting has long been used as a technique concurrently with facial reconstruction procedures and facial rejuvenation procedures as a "filler" of sorts for facial augmentation as early as 1893 (Miller). The fat injected into the face serves as a volume expander to correct defects related to loss of muscle or bone, such as in micrognathia. Since those initial trials, the technique has been widely expanded and honed to provide the best possible contouring. In addition to the filler aspects and results of the procedure, the technique has been observed to improve skin quality in injection sites, improve pigmentation irregularities, and even improve appearance of long standing scars. However, a formal study of fat grafting's potential of improved wound healing and minimization of scar formation has never been undertaken.

Although not identical to the process of injection of autologous ADSCs, the process of fat grafting has the capabilities of providing some number of ADSCs that were in the adipose harvest. Additionally, the process itself has been shown in the past to improve previously existing scars and improve the quality of skin overlying injection sites (Coleman). Therefore, it is logical to assume that injection of autologous fat will improve wound healing and minimize scar formation in patients undergoing the procedure through effects of ADSCs within the harvested tissue.

With the advent of advanced 3-D imaging technology, we are now able to obtain high-quality, high-resolution images to document and detail stages of wound healing and scar formation. Therefore, we will be able to determine through observer analysis whether the process of fat grafting changes the formation and quality of scars over time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects
* Facial reconstruction surgery in the last 3 months

Exclusion Criteria:

* Age less than 18 years
* Patients undergoing skin grafting
* Patients undergoing secondary intent closure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Color, Vascularity, Distortion, Contour, and Appearance of Scar through use of Manchester Scar Scale | 3 months post-fat grafting
  An independent group of observers/evaluators, consisting of medical students and other non-faculty medical personnel as well as general lay observers, will be asked to view the 3-D images from each time point, evaluate the aesthetic outcome, and grade the scars presented in each case. Scales used will be the Manchester Scar Scale, which has been used previously for photographic scar assessment, as well as a more lay-person's version of the Manchester Scar scale created for the use of an average observer. These forms assess the color, hypertrophy, vascularity, etc of the scar as compared to surrounding skin. The data collected will be analyzed using appropriate statistical software and/or calculations.
Color, Vascularity, Distortion, Contour, and Appearance of Scar through use of Manchester Scar Scale | 6 months post-fat grafting
  An independent group of observers/evaluators, consisting of medical students and other non-faculty medical personnel as well as general lay observers, will be asked to view the 3-D images from each time point, evaluate the aesthetic outcome, and grade the scars presented in each case. Scales used will be the Manchester Scar Scale, which has been used previously for photographic scar assessment, as well as a more lay-person's version of the Manchester Scar scale created for the use of an average observer. These forms assess the color, hypertrophy, vascularity, etc of the scar as compared to surrounding skin. The data collected will be analyzed using appropriate statistical software and/or calculations.
Color, Vascularity, Distortion, Contour, and Appearance of Scar through use of Manchester Scar Scale | 12 months post-fat grafting
  An independent group of observers/evaluators, consisting of medical students and other non-faculty medical personnel as well as general lay observers, will be asked to view the 3-D images from each time point, evaluate the aesthetic outcome, and grade the scars presented in each case. Scales used will be the Manchester Scar Scale, which has been used previously for photographic scar assessment, as well as a more lay-person's version of the Manchester Scar scale created for the use of an average observer. These forms assess the color, hypertrophy, vascularity, etc of the scar as compared to surrounding skin. The data collected will be analyzed using appropriate statistical software and/or calculations.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Steinbacher, MD, DMD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

REFERENCES:
- [Background] Soo C, Hu FY, Zhang X, Wang Y, Beanes SR, Lorenz HP, Hedrick MH, Mackool RJ, Plaas A, Kim SJ, Longaker MT, Freymiller E, Ting K. Differential expression of fibromodulin, a transforming growth factor-beta modulator, in fetal skin development and scarless repair. Am J Pathol. 2000 Aug;157(2):423-33. doi: 10.1016/s0002-9440(10)64555-5. PMID 10934147
- [Background] Frantz FW, Bettinger DA, Haynes JH, Johnson DE, Harvey KM, Dalton HP, Yager DR, Diegelmann RF, Cohen IK. Biology of fetal repair: the presence of bacteria in fetal wounds induces an adult-like healing response. J Pediatr Surg. 1993 Mar;28(3):428-33; discussion 433-4. doi: 10.1016/0022-3468(93)90243-e. PMID 8468658
- [Background] Mori R, Shaw TJ, Martin P. Molecular mechanisms linking wound inflammation and fibrosis: knockdown of osteopontin leads to rapid repair and reduced scarring. J Exp Med. 2008 Jan 21;205(1):43-51. doi: 10.1084/jem.20071412. Epub 2008 Jan 7. PMID 18180311
- [Background] Cooper L, Johnson C, Burslem F, Martin P. Wound healing and inflammation genes revealed by array analysis of 'macrophageless' PU.1 null mice. Genome Biol. 2005;6(1):R5. doi: 10.1186/gb-2004-6-1-r5. Epub 2004 Dec 23. PMID 15642097
- [Background] Ebrahimian TG, Pouzoulet F, Squiban C, Buard V, Andre M, Cousin B, Gourmelon P, Benderitter M, Casteilla L, Tamarat R. Cell therapy based on adipose tissue-derived stromal cells promotes physiological and pathological wound healing. Arterioscler Thromb Vasc Biol. 2009 Apr;29(4):503-10. doi: 10.1161/ATVBAHA.108.178962. Epub 2009 Feb 5. PMID 19201690
- [Background] Blanton MW, Hadad I, Johnstone BH, Mund JA, Rogers PI, Eppley BL, March KL. Adipose stromal cells and platelet-rich plasma therapies synergistically increase revascularization during wound healing. Plast Reconstr Surg. 2009 Feb;123(2 Suppl):56S-64S. doi: 10.1097/PRS.0b013e318191be2d. PMID 19182664
- [Background] Yun IS, Jeon YR, Lee WJ, Lee JW, Rah DK, Tark KC, Lew DH. Effect of human adipose derived stem cells on scar formation and remodeling in a pig model: a pilot study. Dermatol Surg. 2012 Oct;38(10):1678-88. doi: 10.1111/j.1524-4725.2012.02495.x. Epub 2012 Jul 16. PMID 22804839
- [Background] Zuk PA, Zhu M, Ashjian P, De Ugarte DA, Huang JI, Mizuno H, Alfonso ZC, Fraser JK, Benhaim P, Hedrick MH. Human adipose tissue is a source of multipotent stem cells. Mol Biol Cell. 2002 Dec;13(12):4279-95. doi: 10.1091/mbc.e02-02-0105. PMID 12475952
- [Background] Miller JJ, Popp JC. Fat hypertrophy after autologous fat transfer. Ophthalmic Plast Reconstr Surg. 2002 May;18(3):228-31. doi: 10.1097/00002341-200205000-00015. PMID 12021657
- [Background] Coleman SR. Structural fat grafting: more than a permanent filler. Plast Reconstr Surg. 2006 Sep;118(3 Suppl):108S-120S. doi: 10.1097/01.prs.0000234610.81672.e7. PMID 16936550
- [Background] Gurtner GC. Wound Healing: Normal and Abnormal. In: Thorne C, Beasley RW, Aston SJ, Bartlett SP, Gurtner GC, Spear SL, eds. Grabb and Smith's Plastic Surgery. Sixth ed: Philadelphia, PA : Lippincott Williams & Wilkins; 2007.